CLINICAL TRIAL: NCT05009043
Title: COVID-19 Vaccine Hesitancy and Perceptions Among Teaching and Assisting Staff at Faculty of Dentistry, Ain Shams University in Egypt: A Cross-Sectional Study.
Brief Title: COVID-19 Vaccine Hesitancy and Dental Faculty Staff Members in Egypt
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mariam Ayman Amin Sharaf (Other)
Responsible Party: Sponsor-Investigator, Mariam Ayman Amin Sharaf, Teaching assistant, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: 960
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Respiratory Infection; Covid19; Vaccine Refusal
Keywords: COVID-19; Healthcare workers; Dentists; Frontline workers; Vaccine acceptance; Vaccine; Vaccine hesitancy
MeSH Terms: conditions — COVID-19; Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Healthcare workers (HCWs) play a vital role in determining the success of vaccination programs. Patient acceptance and vaccination rely greatly on the utilization and attitude of HCWs towards the vaccine, their attitude also influences patients' adherence to vaccination schedules and their hesitancy. HCWs themselves can be hesitant about a certain vaccine and thus can transfer their negative attitudes to their patients, increasing vaccine hesitancy among the general population. Frontline HCWs are at an increased risk of exposure to COVID-19 due to their direct contact with their patients, working hours, psychological stress and job burnout, they also face stigma. Dental health professionals in particular are at an increased risk due to their occupational hazards that include continuous exposure to body fluids and aerosols, this increases their risk of contracting COVID-19. Therefore vaccinating healthcare workers will be beneficial, not only for themselves, but also for their households and patients.

DETAILED DESCRIPTION:
To mitigate the rapid spread of COVID-19 and its massive impact on the economy worldwide, efforts have to be made to protect people against the disease, one of the most effective means was found to be vaccination. The range of technology in the development of COVID-19 vaccine is a striking feature where various approaches are being evaluated including, but not limited to: nucleic acid (DNA and RNA), recombinant protein, live-attenuated virus, inactivated virus and virus-like particles approaches. It is the responsibility of governments to ensure equity in the distribution and access to the novel vaccine. Authorized and currently available vaccines in Egypt include: 1) COVID-19 Vaccine AstraZeneca (AZD1222) which is an adenovirus vaccine manufactured in UK, 2) Sputnik V, a recombinant adenovirus vaccine manufactured in Russia and 3) BBIBP-CorV Sinopharm, which is an inactivated vaccine manufactured in China. The total number of vaccine doses administered in Egypt was reported to be 1,315 doses in March 2021.

However, vaccine availability is not enough to ensure large-scale immunization; success of vaccination programs depend greatly on the population's demand and acceptability of the vaccine. Governments should strive to understand determinants of vaccine acceptability and perception of people towards the vaccine. Although vaccination has largely contributed to decreasing the global burden of diseases and mortality, various factors can affect the acceptance of a new vaccine. "Vaccine hesitancy" has been declared by WHO as one of the ten global health threats worldwide, and has been defined as 'delay in acceptance or refusal of vaccination despite availability of vaccination services.' Causes of vaccine hesitancy include concerns about its safety, efficacy, personal beliefs, religious reasons, concerns about its rapid development as the rapid development of swine flu vaccine was previously associated with increased risk of Guillain-Barre syndrome, low benefits perceived and fear of side effects. Moreover, some people have concerns about the manufacturing process of the vaccine, as a defective polio vaccine lead to development of incident cases of polio and paralysis and death in earlier times.

In Egypt, healthcare workers are the first group to have access to COVID-19 vaccine and hence, act as a primary source of knowledge to the public about the vaccine, therefore it is crucial to estimate their level of perception and acceptability of the vaccine and determine factors affecting their acceptability. This will help inform stakeholders to make decisions regarding COVID-19 vaccination programs. To the best of our knowledge, this is the first study in Egypt targeting dental health professionals in particular, owing to their exclusive high exposure level to COVID-19 among healthcare workers

ELIGIBILITY:
Inclusion Criteria:

* Staff members at Faculty of Dentistry, Ain Shams University
* Egyptians.

Exclusion Criteria:

* Staff members who refuse to participate in the study.
* Staff members currently living abroad. (As their perception about COVID-19 situation and risk in Egypt will not be accurate)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Staff members of Faculty of Dentistry, Ain Shams University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Staff members who accept/refuse vaccination against COVID-19 | August 2021-October 2021
  Percentage

SECONDARY OUTCOMES:
Perceived barriers and enablers of staff members to get vaccinated against COVID-19 | August 2021-December 2021
Factors associated with acceptance of COVID-19 vaccination among staff members. | August 2021-December 2021
  Demographics, previous COVID-19 experience, knowledge and attitude
Risk perception of COVID-19 among staff members. | August 2021-December 2021

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Sharaf, Msc, Principal Investigator — Ain Shams University; Amira Badran, PhD, Study Director — Ain Shams University; Omar Taqa, Msc, Principal Investigator — Ain Shams University; Haneen Zahran, Msc, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No